CLINICAL TRIAL: NCT00687739
Title: Estrogen Deficiency and Mechanisms of Fat Accumulation
Brief Title: Prevention of Obesity in Women Via Estradiol Regulation
Acronym: POWER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 06-0512; R01AG018198 (NIH)
Record Dates: First submitted 2008-05-29; First posted 2008-06-02 (Estimated); Results first posted 2019-12-09 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Obesity
Keywords: hormone therapy; obesity; postmenopause; disease /disorder proneness /risk; insulin sensitivity /resistance; metabolic syndrome; women's health
MeSH Terms: conditions — Obesity; Disease Susceptibility; Metabolic Syndrome | interventions — Leuprolide; Estradiol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Placebo Comparator): GnRH agonist + placebo
  Interventions: Drug: leuprolide acetate
- 2 (Active Comparator): GnRH agonist + placebo + exercise
  Interventions: Drug: leuprolide acetate; Behavioral: progressive resistance exercise training
- 3 (Experimental): GnRH agonist + Estradiol
  Interventions: Drug: leuprolide acetate; Drug: Estradiol Transdermal
- 4 (Experimental): GnRH agonist + Estradiol + exercise
  Interventions: Drug: leuprolide acetate; Drug: Estradiol Transdermal; Behavioral: progressive resistance exercise training

INTERVENTIONS:
Drug: leuprolide acetate — 3.75 mg for depot suspension delivered by monthly intramuscular injection for 5 months
  Other Names: Lupron
Drug: Estradiol Transdermal — 0.075 mg patch per day for 5 months
  Other Names: Climara
  Arms: 3; 4
Behavioral: progressive resistance exercise training — 45 minute exercise sessions 4 times per week for 5 months
  Arms: 2; 4

SUMMARY:
The purpose of this study is to evaluate potential mechanisms by which estradiol deficiency accelerates fat gain and abdominal fat accumulation in women.

DETAILED DESCRIPTION:
Many factors contribute to the current epidemic of obesity. Although estrogen status is not commonly recognized as a determinant of obesity risk in women, there is strong evidence from large randomized controlled trials that estradiol (E2)-based hormone therapy (HT) reduces weight gain by about 40% in postmenopausal women. Importantly, there is also strong evidence that E2 reduces abdominal fat accumulation, a fundamental component of the Metabolic Syndrome. Some studies suggest risks of HT outweigh the benefits for some women. However, this does not negate the importance of learning the mechanisms by which E2 influences energy balance and fat patterning.

This study uses gonadotropin releasing hormone (GnRH) analog therapy to determine the effects of chronic (5-month) sex hormone suppression on resting energy expenditure (REE), altered hypothalamic-pituitary-adrenal (HPA) axis activity, and fat gain.

It is hypothesized that REE will be reduced in response to chronic sex hormone suppression, promoting fat gain. It is also hypothesized that stress-induced hypothalamic-pituitary-adrenal (HPA)axis activity will be amplified during sex hormone suppression; altered HPA axis activity leading to cortisol excess causes abdominal fat accumulation. Finally, it is hypothesized that E2 add-back therapy will lessen these responses.

Participants will be randomized so that half of the women in each treatment arm will participate in an exercise training program, consisting of progressive resistance exercise to prevent the decline in fat-free mass (FFM) and the increase in fat mass that has been observed in young women in response to GnRH analog therapy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy premenopausal women, aged 18 to 49 years
* Regular menses (no missed cycles in previous year; cycle length 25-35 days)
* Positive luteinizing hormone test or a mid-luteal serum progesterone greater than 3 ng/mL
* Nonsmokers
* Willing to receive all study interventions
* Physically able and willing to be randomized to participate in a supervised resistance exercise training program

Exclusion Criteria:

* Already performing high-intensity resistance exercise training more than 1 day per week
* On diabetes medications
* Use of hormonal contraception in the past 3 months
* On oral or inhaled glucocorticoids
* Positive pregnancy test
* Intention to become pregnant or start hormonal contraceptive therapy during the period of study
* Lactation
* Hypersensitivity to extrinsic peptide hormones, mannitol, Gonadotropin-releasing hormone (GnRH), leuprolide acetate, benzyl alcohol (the vehicle for injection of leuprolide acetate), or transdermal patch
* Score greater than 16 on the Center for Epidemiologic Studies Depression Scale and Beck Depression Inventory-II score greater than 18, or clinician recommendation to exclude
* Severe osteopenia or osteoporosis (proximal femur or lumbar spine t scores < -2.0)
* BMI greater than 40 kg/m2, weight change of more than ± 2 kg in last 6 months, or weight-reduced by more than 5 kg from maximal body weight
* Abnormal vaginal bleeding
* History of breast cancer or other estrogen-dependent neoplasms
* History of venous thromboembolic events
* Moderate or severe renal impairment (creatinine clearance <50 mL/min by Cockcroft-Gault)
* Chronic hepatobiliary disease, defined as liver function tests (AST, ALT, alkaline phosphatase, total bilirubin) greater than 1.5 times the upper limit of normal
* Thyroid dysfunction, defined as ultra sensitive TSH less than 0.5 or greater than 5.0 mU/L
* Uncontrolled hypertension, defined as resting BP greater than 150/90 mmHg
* Cardiovascular disease, including indicators of ischemic heart disease or serious arrhythmias at rest or during the graded exercise test; follow-up diagnostic testing to rule out cardiovascular disease by a cardiologist will be allowed
* Orthopedic or other problems that would interfere with participation in the exercise program

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2008-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy M Kohrt, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Background] Anderson GL, Limacher M, Assaf AR, Bassford T, Beresford SA, Black H, Bonds D, Brunner R, Brzyski R, Caan B, Chlebowski R, Curb D, Gass M, Hays J, Heiss G, Hendrix S, Howard BV, Hsia J, Hubbell A, Jackson R, Johnson KC, Judd H, Kotchen JM, Kuller L, LaCroix AZ, Lane D, Langer RD, Lasser N, Lewis CE, Manson J, Margolis K, Ockene J, O'Sullivan MJ, Phillips L, Prentice RL, Ritenbaugh C, Robbins J, Rossouw JE, Sarto G, Stefanick ML, Van Horn L, Wactawski-Wende J, Wallace R, Wassertheil-Smoller S; Women's Health Initiative Steering Committee. Effects of conjugated equine estrogen in postmenopausal women with hysterectomy: the Women's Health Initiative randomized controlled trial. JAMA. 2004 Apr 14;291(14):1701-12. doi: 10.1001/jama.291.14.1701. PMID 15082697
- [Background] Sites CK, L'Hommedieu GD, Toth MJ, Brochu M, Cooper BC, Fairhurst PA. The effect of hormone replacement therapy on body composition, body fat distribution, and insulin sensitivity in menopausal women: a randomized, double-blind, placebo-controlled trial. J Clin Endocrinol Metab. 2005 May;90(5):2701-7. doi: 10.1210/jc.2004-1479. Epub 2005 Feb 1. PMID 15687338
- [Background] Utian WH, Gass ML, Pickar JH. Body mass index does not influence response to treatment, nor does body weight change with lower doses of conjugated estrogens and medroxyprogesterone acetate in early postmenopausal women. Menopause. 2004 May-Jun;11(3):306-14. doi: 10.1097/01.gme.0000117062.54779.bd. PMID 15167310
- [Derived] Gavin KM, Shea KL, Gibbons E, Wolfe P, Schwartz RS, Wierman ME, Kohrt WM. Gonadotropin-releasing hormone agonist in premenopausal women does not alter hypothalamic-pituitary-adrenal axis response to corticotropin-releasing hormone. Am J Physiol Endocrinol Metab. 2018 Aug 1;315(2):E316-E325. doi: 10.1152/ajpendo.00221.2017. Epub 2018 Apr 6. PMID 29631362

RESULTS

PARTICIPANT FLOW:
Groups:
- GnRH Agonist + Placebo: GnRH agonist + placebo
  leuprolide acetate: 3.75 mg for depot suspension delivered by monthly intramuscular injection for 5 months
- GnRH Agonist + Placebo + Exercise: GnRH agonist + placebo + exercise
  leuprolide acetate: 3.75 mg for depot suspension delivered by monthly intramuscular injection for 5 months
  progressive resistance exercise training: 45 minute exercise sessions 4 times per week for 5 months
- GnRH Agonist + Estradiol: GnRH agonist + Estradiol
  leuprolide acetate: 3.75 mg for depot suspension delivered by monthly intramuscular injection for 5 months
  Estradiol Transdermal: 0.075 mg patch per day for 5 months
- GnRH Agonist + Estradiol + Exercise: GnRH agonist + Estradiol + exercise
  leuprolide acetate: 3.75 mg for depot suspension delivered by monthly intramuscular injection for 5 months
  Estradiol Transdermal: 0.075 mg patch per day for 5 months
  progressive resistance exercise training: 45 minute exercise sessions 4 times per week for 5 months
Period: Overall Study
Arm/Group | GnRH Agonist + Placebo | GnRH Agonist + Placebo + Exercise | GnRH Agonist + Estradiol | GnRH Agonist + Estradiol + Exercise
Started | 25 | 15 | 25 | 14
Completed | 23 | 12 | 23 | 12
Not Completed | 2 | 3 | 2 | 2
Not completed — Lost to Follow-up | 2 | 2 | 1 | 2
Not completed — Adverse Event | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Of the 79 women enrolled, 9 discontinued. Baseline and outcome measure data are reported for the 70 participants who completed the study. Ethnic data (Hispanic or Latino) are not distinct from racial data. 9 women who identified as Hispanic or Latino are also included in one of the race categories
Groups:
- Total: Total of all reporting groups
Arm/Group | GnRH Agonist + Placebo | GnRH Agonist + Placebo + Exercise | GnRH Agonist + Estradiol | GnRH Agonist + Estradiol + Exercise | Total
Number analyzed (Participants) | 23 | 12 | 23 | 12 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (8) | 36 (8) | 35 (9) | 35 (9) | 35.5 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 12 | 23 | 12 | 70
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 0 | 0 | 2
  Native American | 1 | 0 | 0 | 0 | 1
  Black | 2 | 1 | 4 | 2 | 9
  Caucasian | 15 | 9 | 17 | 9 | 50
  More than one race | 4 | 1 | 0 | 1 | 6
  Refused to answer | 0 | 0 | 2 | 0 | 2
  Hispanic or Latino | 4 | 2 | 1 | 2 | 9
Region of Enrollment [Number; unit: participants]
  United States | 23 | 12 | 23 | 12 | 70
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28 (6) | 28 (6) | 28 (6) | 28 (6) | 28 (6)
Body Composition Total Mass [Mean (Standard Deviation); unit: kilograms] | 74.4 (2.7) | 74.4 (2.7) | 76.6 (3) | 76.6 (3) | 75.5 (2.8)
Body Composition Fat Mass [Mean (Standard Deviation); unit: kilograms] | 27.8 (1.9) | 27.8 (1.9) | 28.2 (2) | 28.2 (2) | 28 (2)

OUTCOME MEASURES:

1. Primary Outcome: Resting Energy Expenditure (REE)
Description: Resting energy expenditure measured by indirect calorimeter at baseline and after 5 months of treatment.
Time Frame: Before and after 5 months of treatment
Population: Participants who completed 24-h visits in the room calorimeter before and after the intervention. This could not be accomplished in all participants in the trial because of scheduling difficulties and/or lack of availability of the calorimeter. The primary analysis was by drug group only (placebo vs estradiol), collapsed across exercise grouping.
Measure: Mean (95% Confidence Interval); unit: kcal/d
Groups:
- GnRHag+PL: GnRH agonist + placebo
  leuprolide acetate: 3.75 mg for depot suspension delivered by monthly intramuscular injection for 5 months
- GnRHag+PL+ex: GnRH agonist + placebo + exercise
  leuprolide acetate: 3.75 mg for depot suspension delivered by monthly intramuscular injection for 5 months
  progressive resistance exercise training: 45 minute exercise sessions 4 times per week for 5 months
- GnRHag+E2: GnRH agonist + Estradiol
  leuprolide acetate: 3.75 mg for depot suspension delivered by monthly intramuscular injection for 5 months
  Estradiol Transdermal: 0.075 mg patch per day for 5 months
- GnRHag+E2+ex: GnRH agonist + Estradiol + exercise
  leuprolide acetate: 3.75 mg for depot suspension delivered by monthly intramuscular injection for 5 months
  Estradiol Transdermal: 0.075 mg patch per day for 5 months
  progressive resistance exercise training: 45 minute exercise sessions 4 times per week for 5 months
Arm/Group | GnRHag+PL | GnRHag+PL+ex | GnRHag+E2 | GnRHag+E2+ex
Number analyzed (Participants) | 16 | 8 | 16 | 8
kcal/d | -37.8 [-88.7 to 13.0] | -87.2 [-185.9 to 11.4] | 14.6 [-34.8 to 64.0] | -19.3 [-95.1 to 56.4]
Statistical Analysis 1: Comparison: GnRHag+PL vs GnRHag+PL+ex vs GnRHag+E2 vs GnRHag+E2+ex; The primary analysis was the effect of PL vs E2 collapsed across exercise (2-group comparison). The analysis of effects of exercise was exploratory (evaluated within-group changes only); Test type: Superiority — The primary analysis compared the GnRHAG + E2 and GnRHAG + PL groups, pooled across exercise status. It was acknowledged that the inclusion of exercisers could minimize the effects of GnRHAG but would be reflective of the effects of ovarian hormone suppression on sedentary and active women. Differences in changes across time between groups were tested using an analysis of covariance model conditioned on baseline; p < 0.05, ANCOVA — The p value was calculated

2. Primary Outcome: Cortisol Response (Area Under the Curve) to CRH Under DEX Suppression
Description: Cortisol response to corticotropin releasing hormone (CRH) during dexamethasone (DEX) suppression; DEX/CRH stimulation test
Time Frame: Before and after 5 months of treatment
Population: Women who completed the DEX/CRH stimulation test before and after the intervention. The Outcome Measure evaluation was only conducted in a subgroup of women - those in the Drug intervention arms. This evaluation was not done in the exercise arms.
Measure: Mean (95% Confidence Interval); unit: ng/mL x min
Groups:
- GnRHag+E2: GnRH agonist + estradiol
  euprolide acetate: 3.75 mg for depot suspension delivered by monthly intramuscular injection for 5 months
  Estradiol Transdermal: 0.075 mg patch per day for 5 months
Arm/Group | GnRHag+PL | GnRHag+E2
Number analyzed (Participants) | 15 | 15
ng/mL x min | 189 [-2481 to 2859] | -3115 [-5322 to -907]
Statistical Analysis 1: Comparison: GnRHag+PL vs GnRHag+E2; The primary analysis was the comparison of within-group changes in the E2 and placebo groups for cortisol AUC in response to Dex/CRH and between-group differences in the changes. Within-group changes and between-group differences in changes were evaluated by linear contrast using an ANCOVA model with adjustment for pre-intervention values of outcomes; Test type: Superiority; p < 0.05, ANCOVA — The p value was calculated

3. Secondary Outcome: Total Energy Expenditure (TEE)
Description: 24-hour energy expenditure measured by indirect calorimetry in a room calorimeter
Time Frame: Before and after 5 months of treatment
Population: Participants who completed 24-h visits in the room calorimeter before and after the intervention
Measure: Mean (95% Confidence Interval); unit: kcal/d
Arm/Group | GnRHag+PL | GnRHag+PL+ex | GnRHag+E2 | GnRHag+E2+Ex
Number analyzed (Participants) | 16 | 8 | 16 | 8
kcal/d | -108.8 [-201.1 to -16.5] | -166.5 [-388.1 to 55.1] | -92.7 [-167.1 to -18.4] | -107.4 [-298.3 to 83.5]
Statistical Analysis 1: Comparison: GnRHag+PL vs GnRHag+PL+ex vs GnRHag+E2 vs GnRHag+E2+Ex; The primary analysis compared the GnRHag+E2 and GnRHag+PL groups, pooled across exercise status. Differences in change over time between groups were tested by using an ANCOVA model, first with treatment group alone, and again adding FM and FFM to the model; Test type: Superiority; p < 0.05, ANCOVA — The p value was calculated

4. Secondary Outcome: Fat Mass
Description: Total body fat mass measured by DXA
Time Frame: Before and after 5 months of treatment
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | GnRHag+PL | GnRHag+PL+ex | GnRHag+E2 | GnRHag+E2+ex
Number analyzed (Participants) | 23 | 12 | 23 | 12
kg | 0.5 [-0.5 to 1.4] | -0.6 [-1.7 to 0.5] | 0.4 [-0.7 to 1.5] | -0.8 [-2.9 to 1.2]

5. Secondary Outcome: Fat-free Mass
Description: Total body fat-free mass measured by DXA
Time Frame: Before and after 5 months of treatment
Population: Participants who completed outcome measurements before and after the interention
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | GnRHag+PL | GnRHag+PL+ex | GnRHag+E2 | GnRHag+E2+ex
Number analyzed (Participants) | 23 | 12 | 23 | 12
kg | -1.0 [-1.5 to -0.6] | 0.1 [-0.6 to 0.7] | 0.0 [-0.5 to 0.4] | 1.0 [-0.3 to 2.2]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time eligibility was established through the completion of the study, over approximately 1 year.
Description: Adverse events were queried every 4 weeks.
Arm/Group | GnRH Agonist + Placebo | GnRH Agonist + Placebo + Exercise | GnRH Agonist + Estradiol | GnRH Agonist + Estradiol + Exercise
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/12 | 1/23 | 0/12
Other Adverse Events (participants affected / at risk) | 0/23 | 0/12 | 0/23 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GnRH Agonist + Placebo (N=23) | GnRH Agonist + Placebo + Exercise (N=12) | GnRH Agonist + Estradiol (N=23) | GnRH Agonist + Estradiol + Exercise (N=12)
Hospitalization (Product Issues) | 0 | 0 | 1 (1) | 0 — Breast implant ruptured

LIMITATIONS AND CAVEATS:
This was a mechanistically driven study to isolate the effects of estradiol on bioenergetics and HPA axis activity. It was not a therapeutic clinical trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No